CLINICAL TRIAL: NCT02520154
Title: Matched Paired Pharmacodynamics and Feasibility Study of Pembrolizumab in Combination With Chemotherapy in Frontline Ovarian Cancer
Brief Title: Pembrolizumab, Carboplatin, and Paclitaxel in Treating Patients With Stage III-IV Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0662; NCI-2015-01508 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0662 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Results first posted 2024-08-29 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (carboplatin, paclitaxel, and pembrolizumab) (Experimental): NACT: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15, and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  ADJUVANT THERAPY: Beginning 3-6 weeks after surgery, paclitaxel IV over 1 hour on days 1, 8, and 15, patients receive carboplatin IV over 1 hour on day 1, and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 20 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Pembrolizumab; Other: Pharmacological Study

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well pembrolizumab works when given in combination with carboplatin and paclitaxel in treating patients with stage III-IV ovarian, primary peritoneal, or fallopian tube cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab in combination with carboplatin and paclitaxel may be a better treatment for ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate progression-free survival of paclitaxel/carboplatin and pembrolizumab in patients with advanced stage, metastatic ovarian cancer undergoing neoadjuvant chemotherapy (NACT).

SECONDARY OBJECTIVES:

I. To describe the feasibility of combination therapy with pembrolizumab in this population.

II. To evaluate the safety of combination and maintenance pembrolizumab. III. To report overall survival.

EXPLORATORY OBJECTIVES:

I. To describe the sequential effects of chemotherapy on immune response and PD-1 expression and receptor occupancy.

II. To evaluate circulating lymphoid populations (subsets). III. To determine tissue PD-L1 expression and T-cell infiltration.

OUTLINE:

NACT: Patients receive paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15, and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

ADJUVANT THERAPY: Beginning 3-6 weeks after surgery, paclitaxel IV over 1 hour on days 1, 8, and 15, patients receive carboplatin IV over 1 hour on day 1, and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 20 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent
* Histology showing high-grade epithelial non-mucinous ovarian, primary peritoneal, or fallopian tube cancer
* No more than 4 prior cycles of chemotherapy for primary advanced (stage III or IV) epithelial ovarian, primary peritoneal, or fallopian tube cancer
* No prior treatment involving irradiation, hormonal therapy, immunotherapy, investigational therapy, and/or other concurrent agents or therapies for ovarian cancer
* A disposition to neoadjuvant chemotherapy with planned interval tumor reductive surgery after 4 complete cycles of treatment
* Planned dose-dense chemotherapy with combination carboplatin and paclitaxel given intravenously
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

  * Measurable disease is defined at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each "target" lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT
  * Patients with non-measurable but evaluable solid tumors may be deemed eligible contingent upon principal investigator (PI) review
* Peripheral neuropathy grade 0 or 1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
* Tissue from an archival tissue sample or fresh tissue obtained from a core or excisional biopsy of a tumor lesion
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000/mcL
* Hemoglobin (Hgb) >= 9 g/dL or >= 5.6 mmol/L
* Creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 x institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases
* International normalized ratio (INR)/prothrombin time (PT) =< 1.5 x ULN (unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time [PTT] is within therapeutic range of intended use of anticoagulants)
* PTT =< 1.5 x ULN (unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
* Women of child-bearing potential (intact uterus) should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Pre-treatment fresh frozen tissue available for research purposes; this tissue can be collected from preoperative laparoscopy, other diagnostic biopsy, or a research-specific biopsy
* Signed informed consent on protocol LAB02-188

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Histology showing mucinous or low grade epithelial ovarian carcinoma
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and or low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
  * Concomitant stage 1A/B, grade 1-2 endometrioid endometrial cancer as allowable contemporary tumor
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Patients with ovarian cancer not medically fit for diagnostic laparoscopy prior to initiation of therapy
* Patients with any evidence of severe or uncontrolled systemic disease (e.g. severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease], uncontrolled chronic renal disease [glomerulonephritis, nephritic syndrome, Fanconi syndrome or renal tubular acidosis]), or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension blood pressure >= 140/90, active bleeding diatheses or active infection
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study; Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* No active autoimmune disease that has required systemic treatment in past two years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Patients with tuberculosis
* Patients with known hypersensitivity to pembrolizumab or any of its excipients
* Patients receiving concurrent additional biologic therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin, paclitaxel not responsive to traditional desensitization procedures
* Patient that is not able to understand or to comply with the study instructions and requirements or has a history of non-compliance to the medical regimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Jazaeri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] How JA, Dang M, Lee S, Fellman B, Westin SN, Sood AK, Fleming ND, Shafer A, Yuan Y, Liu J, Zhao L, Celestino J, Hajek R, Morgan MB, Parra ER, Laberiano Fernandez CD, Arrechedera CA, Solis Soto LM, Schmeler KM, Nick A, Lu KH, Coleman R, Wang L, Jazaeri AA. Pembrolizumab plus chemotherapy in frontline treatment of advanced ovarian cancer: Clinical and translational results from a phase 2 trial. Med. 2025 Jan 10;6(1):100494. doi: 10.1016/j.medj.2024.07.022. Epub 2024 Aug 15. PMID 39151421
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 07/05/2016 and closed to new patient entry on 09/09/2020. All recruitments were done in a medical clinic setting
Pre-assignment Details: There were 58 participants who were screened for the protocol study. 27 participants were found to be screen failures, 2 participants withdrew from the study, 2 participants were taken off study due to medical concerns by their primary physician, and 1 participants expired from early progression of disease not related to the study treatment. 26 participants were able to complete the study treatments as outlined in the study design
Groups:
- Treatment Group: Paclitaxel 80 mg/m2 IV on Day 1, 8, 15 + Carboplatin AUC of 6 IV on Day 1 for 3 cycles every 21 days, followed by interval debulking surgery, then followed by Pembrolizumab 200 mg IV on Day 1 + Paclitaxel 80 mg/m2 IV on Day 1, 8, 15 + Carboplatin AUC of 6 IV on Day 1 for 3 cycles every 21 days, followed by Pembrolizumab maintenance at 200 mg IV every 21 days for up to 20 additional cycles
Period: Overall Study
Arm/Group | Treatment Group
Started | 31
Completed | 26
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 14
Age, Continuous [Mean (Full Range); unit: years] | 61 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 31
Treatment Group [Count of Participants; unit: Participants] | 31

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Progression-free Survival of Paclitaxel/Carboplatin and Pembrolizumab in Patients With Advanced Stage, Metastatic Ovarian Cancer Undergoing NACT
Description: PFS was defined from the start of neoadjuvant therapy until the date of disease progression or death, whichever occurred first. Disease progression was evaluated using RECIST v1.1 guidelines. Patients who were alive without disease progression were censored at their last evaluation date or until withdrawal of consent. Patients who were removed off protocol for reasons other than disease progression, death, treatment toxicity, or withdrawal of consent were censored at the start date of their non-protocol treatment. Feasibility was defined as the ability to complete all planned 3 cycles of adjuvant carboplatin, paclitaxel, and pembrolizumab.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Group
Number analyzed (Participants) | 31
months | 14.2 [10.5 to 23]

2. Secondary Outcome: To Describe the Feasibility of Combination Therapy and Maintenance Pembrolizumab in This Population
Description: Pembrolizumab with chemotherapy was feasible and resulted in PFS within the historical range for this EOC population.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 31
Participants | 26

3. Secondary Outcome: To Evaluate the Safety of Combination and Maintenance Pembrolizumab
Description: Toxicity was evaluated via grading and recording treatment-related adverse events (TRAE) according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 31
Participants | 31

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: The study was activated on 05/16/2016 and the first patient was registered on study 09/02/2016. The last patient treated on study was taken off treatment on 05/28/2021. Adverse events were reported from baseline till 30 days following the last dose of study agent given.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 13/31
Other Adverse Events (participants affected / at risk) | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=31)
Neutrophil count decrease (Investigations) | 5 (6)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
SGPT increased (Investigations) | 1 (1)
SGOT increased (Investigations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lipid increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=31)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
SGPT increased (Investigations) | 9 (19)
Alk Phos increased (Investigations) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 26 (92)
Anorexia (Metabolism and nutrition disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (16)
SGOT increased (Investigations) | 8 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (2)
MCV decreased (Blood and lymphatic system disorders) | 1 (1)
Enlarged lymph node (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Conjunctivitis (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (11)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema limbs (General disorders) | 1 (1)
T3 level decreased (General disorders) | 1 (1)
T4 level decreased (General disorders) | 1 (1)
TSH level decreased (General disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 8 (14)
Fever (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperthyroidism (General disorders) | 4 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 17 (33)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (General disorders) | 5 (5)
Insomnia (General disorders) | 2 (2)
Lipase increased (Investigations) | 4 (15)
Localized edema (General disorders) | 1 (1)
Increased phosphorus (Metabolism and nutrition disorders) | 3 (6)
LDH increased (Metabolism and nutrition disorders) | 1 (1)
Chloride decreased (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (14)
Neck edema (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 24 (99)
Nystagmus (Nervous system disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (11)
Phlebitis (Vascular disorders) | 1 (1)
Platelet count decreased (Investigations) | 14 (45)
Presyncope (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (9)
Increased BUN (Renal and urinary disorders) | 2 (2)
Increased leukocytes in urine (Renal and urinary disorders) | 1 (1)
Nasal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 5 (8)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Tinnitus (General disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal dryness (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
White blood count decreased (Investigations) | 25 (99)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02520154/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT02520154/ICF_001.pdf